CLINICAL TRIAL: NCT03740932
Title: Biomechanical Changes in Women With Post-partum Pelvic Girdle Pain
Brief Title: Biomechanical Changes in Women With Chronic Pelvic Pain
Acronym: biomechanical
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, Doctor, Misr University for Science and Technology
Other Study IDs: P.T.REC/012/001887
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group (group A):: It will consist of 30 subjects who will have cyclic pelvic pain
  Interventions: Diagnostic Test: Study group (group A)
- Study group (group B):: It will consist of 30 subjects who will have non cyclic pelvic pain.
  Interventions: Diagnostic Test: Study group (group A)
- Control group (group C):: It will consist of 30 subjects normal women who will not having pelvic pain.
  Interventions: Diagnostic Test: Study group (group A)

INTERVENTIONS:
Diagnostic Test: Study group (group A) — Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimetres, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure

SUMMARY:
Chronic pelvic pain (CPP), a frequent complaint in clinical gynaecology, is defined as cyclic or acyclic pain located in the pelvis, persisting for 6 months or more, and severe enough to cause functional incapacity that requires medical or surgical treatment (or both). Chronic pelvic pain is the reason for approximately 10% of all gynaecologic consultations

DETAILED DESCRIPTION:
Women who showed an imbalance of the pelvis also experienced greater pain. A possible explanation for this is that the change in the position of the uterus, due to the imbalance of the pelvis, prompted an excessive amount of prostaglandin to be secreted. When the spinal alignment of women who had intense menstrual pain was put back to normal, the pain was alleviated. The level of tension in the ligaments and nerves connecting the sacral vertebrae and the uterus is the cause off the menstrual pain. Due to the abnormal restriction of movement of the lumbosacral vertebrae, body fluid increase within the pelvis as wells contraction of the uterus leading to the intensification of the menstrual pain.

Stabilization of anterior and lateral pelvic curves through exercise or osteopathic manipulative techniques that utilizes techniques of muscle energy, balanced ligamentous tension, myofascial release, strain and counterstrain to assist muscles to keep the spine upright and sufficiently flexible to support good posture . Correct posture involves a straight spine, which maintains the natural curve of the spine in the human body. Correct posture minimizes the strain on the human body by maintaining balance of the muscles and skeleton. This balanced musculoskeletal state protects the supporting structures in the body and prevents damage or progressive deformation in all positions, including standing, lying down, and sitting. Additionally, correct posture implies not inclining the body forward, backward, left, or right.

The temporomandibular joint is surrounded by ligaments, muscles, nerves, and blood vessels. The masticatory muscles enable mouth opening and closing, lateral movement, and forward and backward movement of the mouth, and excessive tension or imbalance of muscles can limit the joint movements, possibly resulting in limited ROM. Thus, it can be surmised that the imbalance in the spinal muscles caused the imbalance in the temporomandibular muscles and limited TMJ mobility.

ELIGIBILITY:
Inclusion Criteria:

* The age of the participants will be ranged from 20 to 40 years.
* Their body mass index will be ranged from 20 to 25 kg/m2.
* They will have regular menstrual cycle.
* They will not receive any hormonal therapy or taking any regular drugs.

Exclusion Criteria:

* Bone disease.
* Discogenic state with radiculopathy or not.
* Systemic disease of musculoskeletal system.
* Any sensory problems.
* Previous vertebral fractures.
* Major spinal structural abnormality.
* Major jaw abnormality.
* Any jaw orthotics or prosthesis.
* Missing teeth.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 90 women will participate in this study, thirty women diagnosed as having cyclic pelvic pain and thirty women diagnosed as having non cyclic pelvic pain thirty women normal women will not having pelvic pain. They will be selected from outpatient clinic of obstetrics and Gynaecology department in El-Hosary family health Centre.
  All participants will be given a full explanation of the protocol of the study and informed consent form will be signed from each subject before participating in the study (
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-11 (Actual)

PRIMARY OUTCOMES:
body mass index | 3 months
  BMI in kg/m^2
Satisfaction assessed by the VAS | 3 months
  Degrees of menstrual pain will be assessed using a VAS, which was a method of representing subjects' pain on a 10 cm linear scale. Score of 0 meant 'no pain' and 10 meant 'worst pain'. Tomeasure specific symptoms, such as the s
Pelvic tilt in degrees: | 3 months
  The blocks are released and the rods are placed over the crest of the ilium. The blocks are then pressed firmly toward the midline. Read the angle from the level. If the gauge reads over 21/2°, the result is listed as positive.Anterior pelvic tilting angle: PALM was used for measuring pelvic tilting angle. A mark was put on a point just inferior to ASIS; another mark was put just inferior to PSIS. The callipers of the PALM were put on these two points
jaw movement | 3 months
  Maximal vertical mouth opening (MIO):
  From sitting position, with the use of the calliper, the distance between the incisal edges along the midline of the upper and lower central incisors without pain was measured, by placing one end of the poley gauge against the incisal edge of one of the upper central incisors, and the other end against the incisal edge of the opposing lower incisor.
  The distance recorded in millimeters, the subjects was instructed to" open your mouth as wide as possible without causing pain or discomfort". The poley gauge was sterilized with antiseptic solution before and after each measure
Spinal curves Measurement | 3 months
  spinal inclinations followed standardized procedure. Initially, with the subject in prone lying, reference points were marked at the left and right posterior superior iliac spines (PSIS) and at the intersection of the line joining them over the sacral surface and the vertical line of the spine. Also marked were the interspaces of L5-S1, T12-LI and TI-T2. All measurements of spinal inclinations were taken with the subject in erect standing, with feet together, hands by the sides, head erect and eyes focused directly ahead.For the sagittal curves of the spine, the inclinometer was placed along the slope of the vertebrae at each of the levels of the three marked interspaces, so that the zero reading of the inclinometer matched the marked point. The vertically hanging needle of the inclinometer indicated the angles of inclination of these three levels. From these values, the angles of lordosis and kyphosis were determined

CONTACTS AND LOCATIONS:
Locations (1):
- Rovan Elbesh, Giza, Egypt

REFERENCES:
- [Derived] Kamal EE, Hamada HA, Ashour RS, Yousef AM, Elbesh RM. Biomechanical changes in females with poly cystic ovarian syndrome: a case-control study. Sci Rep. 2025 Apr 1;15(1):11190. doi: 10.1038/s41598-025-93481-9. PMID 40169684